CLINICAL TRIAL: NCT02748278
Title: Comparison of the Number of Oocytes Obtained Between Chinese and Caucasian Women Undergoing in Vitro Fertilization Treatment With a Standard Ovarian Stimulation Regimen
Brief Title: Comparison of the Number of Oocytes Obtained Between Chinese and Caucasian Women in IVF Treatment
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Other Study IDs: UW 15-547
Record Dates: First submitted 2016-04-13; First posted 2016-04-22 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2020-07

CONDITIONS: Subfertility
Keywords: subfertility; In-vitro fertilization
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be saved for genetic study if there is significant difference in the number of oocytes obtained between Chinese and Caucasian women.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Transvaginal ultrasound-guided oocyte retrieval — Transvaginal ultrasound-guided oocyte retrieval will be performed 34-36 hours after hCG injection.
Procedure: Embryo transfer — One or two embryos will be replaced on day 2-5 after oocyte retrieval.

SUMMARY:
IVF is a well-established method to treat various causes of infertility. Some studies have suggested that ethnicity affects the success of IVF. This is a prospective study involving two tertiary IVF units in Hong Kong and Australia. The IVF outcome between Chinese and Caucasians will be compared.

DETAILED DESCRIPTION:
This is a prospective study conducted in two tertiary IVF units in Hong Kong and Australia.

The target population for the trial will be women undergoing IVF or intracytoplasmic sperm injection (ICSI) treatment in two IVF Units.

Intervention:

Patients recruited in this study will undergo IVF+/-ICSI treatment. They will undergo an ultrasound scan on the second or third day (day 2 or 3) of a period to exclude the presence of ovarian cyst and have the antral follicle count determined, which includes all follicles of 2-10 mm measured with a 5.5-7.5mHz transvaginal ultrasound probe. Blood will be checked for anti-mullerian hormone (AMH) measured by Beckman-Coulter Diagnostics.

Ovarian stimulation will be started if there are no ovarian cysts on ultrasound scan. They will receive one long acting gonadotrophin injection Elonva 150 microgram subcutaneously followed by daily gonadotrophin injections (Puregon) 200 IU in an antagonist protocol. Antagonist (orgalutran 0.25 mg) will be started on day 5 of ovarian stimulation. Transvaginal ultrasound will be performed for follicular tracking 7 days after the Elonva injection and every 1-3 days thereafter. No adjustment in FSH dose is allowed. Cycles will be cancelled if there are less than 3 follicles larger than 18mm after one week of 200 IU Puregon or there no developing follicle (i.e. larger than 11mm) after one week of 200 IU Puregon.

Recombinant hCG (Ovidrel, Serono, Bari, Italy) 0.25mg will be given if there are 2 follicles >18 mm in diameter. Gonadotrophin injection will not be given on the day of hCG. Agonist trigger will be used if oestradiol concentration on the day of trigger is greater than 15,000 pmol/L or there are more than 15 follicles >16mm on transvaginal scanning. All embryos or blastocysts will be frozen for transfer later following agonist trigger or when the number of oocytes aspirated is 20 or more. Serum FSH, oestradiol, LH and progesterone concentrations are taken 7 days after the Elonva injection and hCG trigger day. Transvaginal ultrasound-guided oocyte retrieval (TUGOR) will be scheduled on Mondays, Wednesdays and Fridays, 34-36 hours after the hCG injection. Flushing of follicles will not be performed. Follicular fluid not contaminated with blood will be collected from the first and largest follicle on each side for estradiol and progesterone level.

The retrieved oocyte will be inseminated conventionally or by ICSI, depending on the semen parameters. ICSI is advised if the total motile sperm number after sperm preparation < 0.2 million, sperm morphology by strict criteria < 3% or fertilization rate < 30% in previous IVF cycles with conventional insemination. One to two embryos will be replaced on day 2-5 after oocyte retrieval. Luteal phase support will be started according to the standard protocol of the centre. Patients will be followed up for urinary pregnancy test 16 days after embryo transfer. Patients with a positive pregnancy test will have transvaginal ultrasound scan performed 10-14 days later and are referred for antenatal care at 8-10 weeks gestation. The remaining embryos will be frozen. Pregnancy outcome will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-36 years old
* Body weight >60Kg
* Total antral follicle count >=7 and ≤ 20 i.e. not poor ovarian reserve based on Bologna criteria
* Chinese women in the HK centre and Caucasian women (defined as originating from the United Kingdom, Europe or United States of America, excluding the Middle East) in the Australian centre
* Written informed consent

Exclusion Criteria:

* Mixed race/ ethnicity
* History of ovarian surgery
* Body mass index >35 kg/m2
* >2 previous stimulated IVF cycles
* History of ovarian hyperstimulation syndrome in previous stimulated IVF cycles
* Polycystic ovary syndrome or total antral follicle count >20

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing IVF or intracytoplasmic sperm injection (ICSI) treatment in the two study sites.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Number of oocytes obtained | 17 days
  Number of oocytes obtained

SECONDARY OUTCOMES:
Number of follicles smaller than 14, 16mm and larger than 18mm in diameter on day 8 and day of hCG | 8 and day of hCG
  Number of follicles smaller than 14, 16mm and larger than 18mm in diameter on day 8 and day of hCG
Duration of recombinant FSH | 15 days
  Duration of recombinant FSH
Dosage of recombinant FSH | 15 days
  Dosage of recombinant FSH
Serum estradiol levels on day 9 and day of hCG | 9 and day of hCG
  Serum estradiol levels on day 9 and day of hCG
Serum FSH levels on day 9 and day of hCG | 9 and day of hCG
  Serum FSH levels on day 9 and day of hCG
Serum LH levels on day 9 and day of hCG | 9 and day of hCG
  Serum LH levels on day 9 and day of hCG
Serum progesterone levels on day 9 and day of hCG | 9 and day of hCG
  Serum progesterone levels on day 9 and day of hCG
Miscarriage rate | 24 weeks
  Miscarriage rate
Clinical pregnancy rate | 6 weeks
  Clinical pregnancy rate: presence of intrauterine gestational sac at 6 weeks
Ongoing pregnancy rate | 12 weeks
  Ongoing pregnancy rate: presence of fetal heart pulsation on transvaginal scan at 12 weeks
Live birth rate | 44 weeks
  Live birth rate
Ovarian hyperstimulation rate | 8 weeks
  Ovarian hyperstimulation rate (according to RCOG guideline)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest HY Ng, Principal Investigator — Department of Obstetrics and Gynaecology, 6/F, Professorial Block, Queen Mary Hospital, 102 Pokfulam Road, Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ko JKY, Kan A, Leung P, Lee VCY, Li RHW, Ledger W, Ng EHY. Comparison of the number of oocytes obtained after ovarian stimulation between Chinese and Caucasian women undergoing in vitro fertilization using a standardized stimulation regime. J Ovarian Res. 2021 Dec 11;14(1):175. doi: 10.1186/s13048-021-00928-4. PMID 34895264